CLINICAL TRIAL: NCT07166549
Title: A Phase I Trial of Bispecific Anti-CD19, Anti-CD20 CAR T Cells for B Cell Malignancies
Brief Title: Bispecific CAR T Cells for B-cell Malignancies (BaseCAR-01 Trial)
Acronym: BaseCAR-01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01562, th23Holbro
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: B Cell Malignancies; B-cell Leukemia; B Cell Lymphoma; Bispecific Chimeric Antigen Receptor (CAR) T Cells; Relapsed or Refractory (r/r) B-cell Malignancies
Keywords: Bispecific anti-CD19, anti-CD20 CAR T cell therapy; lymphapheresis; lymphodepleting (non- myeloablative) chemotherapy; Immune effector cell-associated neurotoxicity syndrome (ICANS); Cytokine release syndrome (CRS); Immune effector cell-associated haematotoxicity (ICAHT); European Group for Blood and Marrow Transplantation (EBMT); 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG); positron emission computed tomography (PET CT); acute lymphocytic leukemia (ALL); immunoglobulin heavy chain (IGH); non-Hodgkin's lymphoma (NHL); Eastern Cooperative Oncology Group (ECOG)
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell; Recurrence; Cytokine Release Syndrome; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Intervention: Bispecific anti-CD19, anti-CD20 CAR T cells (Experimental): Bispecific anti-CD19, anti-CD20 CAR T cells administration
  Interventions: Drug: Experimental Intervention

INTERVENTIONS:
Drug: Experimental Intervention — The study intervention includes:
  * Lymphapheresis
  * Lymphodepleting chemotherapy
  * CAR-T infusion
  Lymphocytes will be collected from the patients by lymphapheresis to produce a personalized IMP, bispecific anti-CD19, anti-CD20 CAR T cells, which will be manufactured at the GMP facility of the University Hospital Basel.
  Patients receive a preparative lymphodepleting chemotherapy of intravenous cyclophosphamide and fludarabine from day -5 until day -3 (or Bendamustine on day -3 and day -2), before anti-CD19/20 CAR T cells are infused (day 0 = day of infusion).
  Participants will undergo lymphapheresis 2-8 weeks prior to CAR T cell infusion.

SUMMARY:
This study is to provide locally produced, bispecific CD19 CD20 CAR T cells to patients with B-cell lymphoma/leukemia who have no access to commercial CAR T cells or who have relapsed thereafter. The primary objective is to assess the safety of bispecific anti-CD19, anti- CD20 CAR T cell-therapies after lymphodepleting chemotherapy in patients with B cell malignancies with exhausted standard treatment options.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) T cells are engineered T-lymphocytes with artificial receptors, containing domains of a T cell receptor as well as a B cell receptor with predefined specificity to a target antigen. In patients with relapsed or refractory (r/r) B-cell malignancies, who would otherwise have a poor prognosis, CD19-directed CAR T cell therapy showed high response rates. A common cause of relapse is loss of the target antigen on the tumor cells, e.g. CD19. In such cases, further approved treatment options are very limited to date, but recent preclinical and early clinical studies have shown that bispecific anti-CD19, anti-CD20 CAR T cells can overcome this hurdle, adding a second target and leading to excellent outcomes in heavily pretreated patients.

This study is to provide locally produced, bispecific CD19 CD20 CAR T cells to patients with B-cell lymphoma/leukemia who have no access to commercial CAR T cells or who have relapsed thereafter. The primary objective is to assess the safety of bispecific anti-CD19, anti- CD20 CAR T cell-therapies after lymphodepleting chemotherapy in patients with B cell malignancies with exhausted standard treatment options. A secondary objective is the assessment of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of B-cell NHL or B-ALL with relapsed, refractory disease and no available standard therapeutic options (including commercially accessible CAR T products), including:

  * Acute B-lymphoblastic leukaemia
  * Burkitt lymphoma
  * Primary CNS lymphoma
  * DLBCL or high-grade lymphoma of any subtype
  * Primary mediastinal B cell lymphoma (including grey zone lymphoma)
  * Mantle Cell lymphoma
  * Low-grade B-cell NHLs: Follicular lymphoma, chronic lymphocytic leukaemia (CLL)/ small lymphocytic lymphoma (SLL), marginal zone lymphoma, hairy cell leukaemia, splenic B-cell lymphoma/leukaemia with prominent nucleoli, and lymphoplasmacytic lymphoma
* CD19 and/or CD20 positive disease on most recent evaluation (by immunohistochemistry or flow cytometry)
* ECOG clinical performance status ≤2
* Able to provide written informed consent.
* Adequate organ function and bone marrow reserve, unless clearly caused by lymphoma and considered reversible, defined as:

  * Adequate hepatic function: Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤3.0 × (ULN) and serum bilirubin ≤2.0 × ULN (except in congenital hyperbilirubinemia, such as Gilbert syndrome, where direct bilirubin ≤3.0 × ULN is allowed)
  * Adequate renal function: creatinine clearance ≥30 mL/min/1.73 m2
  * Adequate pulmonary function: Forced Expiratory Volume in 1 second (FEV1) ≥50% (with adequate compliance) and pulse oxygenation > 91% with room air.
  * Adequate cardiac function: Left Ventricular Ejection Fraction (LVEF) ≥ 40%, and no clinically significant arrhythmia
  * Adequate bone marrow reserve (Hemoglobin ≥80 g/L (with or without recombinant erythropoietin or red blood cell transfusions), Platelets ≥ 50×10^9/L (with or without platelet transfusions), Absolute Neutrophil Count (ANC) 1.0 ×10^9/L (prior growth factor support is permitted but must be without support in the 7 days before the laboratory test), Absolute Lymphocyte Count ≥0.3 ×10^9/L)
* Willingness to practice highly effective methods of birth control, and, in females of childbearing potential, negative urine or serum pregnancy test before study inclusion, lymphapheresis, and lymphodepleting chemotherapy.

Exclusion Criteria:

* Requirement for systemic corticosteroids, i.e. ≥20 mg of prednisone or equivalent daily. Other immunosuppressive drugs
* Any organ failure, respectively not meeting the inclusion criteria of adequate organ function, or active, BKuncontrolled autoimmune disease.
* Uncontrolled coronary artery disease or uncontrolled arrhythmias
* Stroke within the previous 6 months, a history of neurodegenerative disorder or overt clinical evidence of dementia or altered mental status.
* Seizure within 6 months of signing the ICF unless related to the primary disease (e.g. CNS lymphoma).
* Active secondary malignancy that progressed or required treatment in the last 24 months, other than basal or squamous cell carcinomas of the skin. Further allowed exceptions are: Non-muscle-invasive bladder cancer, non-invasive cervical cancer, or other malignancy that is considered cured or to have a minimal risk of recurrence (e.g. a history of localized prostate or localized and treated breast cancer).
* Uncontrolled active bacterial, fungal, or viral infections, particularly active hepatitis B, hepatitis C, or HIV infection.
* Contraindications, known life-threatening allergies, hypersensitivity, or intolerance to any of the study treatments, including previous severe reactions to dimethyl-sulfoxide
* Cytotoxic chemotherapy within 14 days before apheresis collection for CAR-T cells, respectively 12 weeks for Bendamustin and Fludarabine, and 6 months for Alemtuzumab and ATG.
* Cytotoxic chemotherapy (except for lymphodepletion) within 14 days of CAR-T cell infusion.
* Patients who have undergone allogeneic hematopoietic stem cell transplantation less than 12 weeks ago, have evidence of active graft-versus-host-disease (GVHD) of any grade, or are currently on immunosuppression.
* Previous CAR-T cell therapy within 12 weeks of planned CAR-T cell infusion.
* Investigational treatments within other trials ≤ 4 weeks before enrollment.
* Lack of safe contraception; Women who are pregnant or breastfeeding; and men who plan to father a child while enrolled in this study within 1 year of receiving bispecific anti-CD20, anti-CD19 CAR T cells.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Adverse Events | up to 3 months after CAR T cell infusion
  All adverse events will be assessed in a structured manner (time of onset, duration, resolution, action been taken, assessment of intensity, relationship with study treatment), using the CTCAE Version v5.0.
Evaluation of Adverse Events of special interest (CRS) | up to 3 months after CAR T cell infusion
  All adverse events of special interest (CRS) will be assessed in a structured manner (time of onset, duration, resolution, action been taken, assessment of intensity, relationship with study treatment), using the ASTCT CRS Consensus Grading (Grade 1 up to Grade 4; with Grade 4 as most severe CRS Grade)
Evaluation of Adverse Events of special interest (ICANS) | up to 3 months after CAR T cell infusion
  All adverse events of special interest (ICANS) will be assessed in a structured manner (time of onset, duration, resolution, action been taken, assessment of intensity, relationship with study treatment), using the Immune-effector Cell-associated Encephalopathy (ICE) test, which was developed to provide objectivity for screening and grading the severity of ICANS. The ICE score is performed at least every 8 hours during in-patient care and at every outpatient visit. A higher score indicates better cognitive function, with a perfect score of 10 signifying no impairment.
Evaluation of Adverse Events of special interest (ICAHT) | up to 3 months after CAR T cell infusion
  Evaluation of Adverse Events of special interest (ICAHT) will be assessed in a structured manner (time of onset, duration, resolution, action been taken, assessment of intensity, relationship with study treatment), using the EHA/EBMT consensus grading. The EHA/EBMT consensus grading score is a classification system based on depth and duration of neutropenia.

SECONDARY OUTCOMES:
Objective response rate (ORR): Change in metabolic response in FDG-PET/CT scan | 1, 3, 6 and 12 months after CAR T cell infusion
  For lymphomas and B-cell ALL with lymphadenopathy metabolic response in FDG-PET/CT scan according to the Lugano Classification (Response assessment: Complete Remission; Partial Remission; Progressive Disease)
Objective response rate (ORR): Change in minimal residual disease (MRD) negativity in blood | 1, 3, 6 and 12 months after CAR T cell infusion
  For patients with B-cell ALL minimal residual disease (MRD) negativity as determined by flow cytometry
Objective response rate (ORR): Change in minimal residual disease (MRD) negativity in bone marrow | 1, 3, 6 and 12 months after CAR T cell infusion
  For patients with B-cell ALL minimal residual disease (MRD) negativity as determined by flow cytometry
Objective response rate (ORR): Change in sustained MRD-negative Complete Remission (CR) | 1, 3, 6 and 12 months after CAR T cell infusion
  For patients with B-cell ALL: Sustained MRD-negative CR determined by polymerase chain reaction of the IgH rearrangement
Progression-free survival | up to 12 months after CAR T cell infusion
  Progression-free survival, defined as the time between infusion of CAR T product to progression or death, whichever occurs first
Event free survival | up to 3 months after CAR T cell infusion
  Event free survival, defined as time between infusion of CAR T product to not achieving complete remission 3 months after CAR T infusion, progression, or death, whichever occurs first.
Overall survival | up to 12 months after CAR T cell infusion
  Overall survival, defined as the time between the day of infusion of CAR T product to death of any cause.
Cumulative incidence of non-relapse mortality | up to 12 months after CAR T cell infusion
  Cumulative incidence of non-relapse mortality, defined as any death not related to underlying lymphoid malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Holbro, Prof. Dr., Principal Investigator — University Hospital Basel, Division of Hematology
Locations (1):
- University Hospital Basel, Division of Hematology or Medical Oncology, Basel, Canton of Basel-City, Switzerland